CLINICAL TRIAL: NCT03861403
Title: A Dose Escalation and Expansion Study of TRX518 in Combination With Cyclophosphamide Plus Avelumab in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Product development discontinued unrelated to safety.
Sponsor: Leap Therapeutics, Inc. (Industry)
Collaborators: Pfizer (Industry); Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRX518-004
Record Dates: First submitted 2019-02-26; First posted 2019-03-04 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Solid Tumors; Advanced Triple Negative Breast Cancer; Advanced Hormone Receptor Positive/Endocrine Refractory Breast Cancer; Advanced Metastatic Castration-Resistant Prostate Cancer; Advanced Platinum-Resistant Ovarian Cancer
Keywords: Metastatic; Stage III or IV; Recurrent; Refractory; Solid tumors; Breast cancer; Prostate cancer; Ovarian cancer
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence; Breast Neoplasms; Prostatic Neoplasms; Ovarian Neoplasms | interventions — Cyclophosphamide; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- All Solid Tumors (Experimental): Phase 1b, Part 1 Dose Escalation: TRX518 + CTX Combination (28-Day Cycle):
  Subjects receive the following treatment:
  * Fixed dose of TRX518 administered intravenously on D2 and D16 per cycle
  * Assigned dose of cyclophosphamide administered intravenously on C1D1 and may be re-administered on D1 of a subsequent cycle
  Phase 1b, Part 2 Dose Escalation: TRX518 + CTX + avelumab in (28-Day Cycle):
  Subjects receive the following treatment:
  * Fixed dose of TRX518 administered intravenously on D2 and D16 per cycle
  * Fixed dose of avelumab administered intravenously on D2 and D16 per cycle
  * Fixed dose of cyclophosphamide administered at the MTD from Part 1 intravenously on C1D1 and may be re-administered on D1 of a subsequent cycle
  Interventions: Drug: TRX518; Drug: Cyclophosphamide; Drug: Avelumab
- Advanced Triple Negative Breast Cancer (Experimental): Phase 2a Dose Expansion: TRX518 + CTX Combination + avelumab (28-Day Cycle):
  Subjects receive the following treatment:
  * Fixed dose of TRX518 administered intravenously on D2 and D16 per cycle
  * Fixed dose of avelumab administered intravenously on D2 and D16 per cycle
  * Fixed dose of cyclophosphamide identified in Phase 1b administered on C1D1 and may be re-administered on D1 of a subsequent cycle
  Interventions: Drug: TRX518; Drug: Cyclophosphamide; Drug: Avelumab
- Advanced Hormone Receptor+/Endocrine Refractory Breast Cancer (Experimental): Phase 2a Dose Expansion: TRX518 + CTX Combination + avelumab (28-Day Cycle):
  Subjects receive the following treatment:
  * Fixed dose of TRX518 administered intravenously on D2 and D16 per cycle
  * Fixed dose of avelumab administered intravenously on D2 and D16 per cycle
  * Fixed dose of cyclophosphamide identified in Phase 1b administered on C1D1 and may be re-administered on D1 of a subsequent cycle
  Interventions: Drug: TRX518; Drug: Cyclophosphamide; Drug: Avelumab
- Advanced Metastatic Castration-Resistant Prostate Cancer (Experimental): Phase 2a Dose Expansion: TRX518 + CTX Combination + avelumab (28-Day Cycle):
  Subjects receive the following treatment:
  * Fixed dose of TRX518 administered intravenously on D2 and D16 per cycle
  * Fixed dose of avelumab administered intravenously on D2 and D16 per cycle
  * Fixed dose of cyclophosphamide identified in Phase 1b administered on C1D1 and may be re-administered on D1 of a subsequent cycle
  Interventions: Drug: TRX518; Drug: Cyclophosphamide; Drug: Avelumab
- Advanced Platinum-Resistant Ovarian Cancer (Experimental): Phase 2a Dose Expansion: TRX518 + CTX Combination + avelumab (28-Day Cycle):
  Subjects receive the following treatment:
  * Fixed dose of TRX518 administered intravenously on D2 and D16 per cycle
  * Fixed dose of avelumab administered intravenously on D2 and D16 per cycle
  * Fixed dose of cyclophosphamide identified in Phase 1b administered on C1D1 and may be re-administered on D1 of a subsequent cycle
  Interventions: Drug: TRX518; Drug: Cyclophosphamide; Drug: Avelumab

INTERVENTIONS:
Drug: TRX518 — Administered by IV infusion
Drug: Cyclophosphamide — Administered by IV infusion
Drug: Avelumab — Administered by IV infusion
  Other Names: BAVENCIO®

SUMMARY:
This is a Phase 1b/2a dose escalation and expansion, multi-center study to be conducted in 2 phases:

* Phase 1b

  * Dose Escalation Part 1 (Doublet Therapy)
  * Dose Escalation Part 2 (Triplet Therapy)
* Phase 2a

  * Dose Expansion (Triplet Therapy)

Approximately 125 adult patients with histologically confirmed advanced solid tumors requiring therapy will be enrolled in the study. It is expected that approximately 24 patients will be enrolled in up to 4 cohorts, 2 cohorts in Dose Escalation Part 1 and 2 cohorts in Dose Escalation Part 2, of up to 6 patients per cohort. Up to 98 additional patients will be enrolled in the Dose Expansion phase of the study to achieve 88 evaluable patients (i.e., received at least 1 dose of study drug(s) and have 1 evaluable post-baseline modified RECIST v1.1 tumor response assessment; for mCRPC, assessment of soft tissue response will be per modified RECIST v1.1 and bone progression assessment will be per PCWG3 guidelines or discontinued treatment due to death, toxicity, or clinical progression) over 4 independent expansion groups.In either phase (1b or 2a), patients discontinuing for reasons unrelated to study treatment toxicity prior to completion of Cycle (C) 1 may be replaced to achieve the number of required evaluable patients per cancer type following consultation with the Sponsor. Data from each cohort in the Dose Escalation phase will be evaluated independently for safety and dose limiting toxicities (DLTs) prior to dose escalation and again prior to the Dose Expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Solid Malignancies in Dose Escalation Parts 1 and 2:

  * Histologically documented metastatic or locally advanced, incurable solid malignancy.
  * At least one prior line of systemic therapy for metastatic or locally advanced disease.
* Advanced Triple Negative Breast Cancer (Dose Expansion):

  * Histologically proven invasive breast carcinoma with triple-negative receptor status.
  * At least 1 but no more than 2 prior lines of chemotherapy for metastatic or locally advanced disease.
* Advanced Hormone Receptor-Positive/Endocrine-Refractory Breast Cancer (Dose Expansion):

  * Histologically proven invasive breast carcinoma with hormone receptor+, HER2- status.
  * Only postmenopausal women are eligible. - Previously received at least 1 line of aromatase inhibitor ± cyclin dependent kinase 4 and 6 (CDK4/6) inhibitor therapy. Prior combination therapies of AI or selective estrogen receptor degrader (SERD [fulvestrant]) ± CDK 4/6 inhibitor or AI plus everolimus will be permitted. Up to 1 prior line of systemic chemotherapy for metastatic disease is allowed.
* Advanced Metastatic Castration-Resistant Prostate Cancer (Dose Expansion):

  * Histologically or cytologically confirmed prostate adenocarcinoma or poorly differentiated carcinoma of the prostate.
  * Surgically or medically castrated, with testosterone levels of < 50 ng/dL (< 2.0 nM). If a patient is being treated with LHRH agonists, this therapy must have been initiated at least 4 weeks prior to treatment start and must be continued throughout the study.
  * Patients must have received ≥1 androgen receptor (AR) signaling inhibitors and had disease progression RECIST v1.1 after no more than 1 prior chemotherapy for mCRPC.
* Advanced Platinum-Resistant Ovarian Cancer (Dose Expansion):

  * Histologically or cytologically confirmed diagnosis of metastatic, advanced, or recurrent platinum-resistant epithelial ovarian, primary peritoneal or fallopian tube cancer.
  * Platinum-resistant ovarian cancer defined as disease progression following a response within 180 days following the last administered dose of platinum therapy. Patients who have lack of response (SD) or disease progression while receiving the most recent platinum-based therapy are not eligible.
  * Received up to 3 lines of systemic therapy for platinum-sensitive disease, with the most recent regimen platinum-containing, and no prior systemic therapy for platinum-resistant or refractory disease.
* General:

  * Tumor tissue for mandatory pre-treatment and on-treatment biopsies.
  * One or more tumors measurable on radiographic imaging defined by RECIST 1.1.
  * Adult patients ≥18 years of age.
  * ECOG performance status (PS) score of 0 or 1.
  * Life expectancy of at least 12 weeks.
  * Disease-free of active second/secondary or prior malignancies for ≥2 years, with the exception of currently treated basal cell or squamous cell carcinoma of the skin or carcinoma in-situ of the cervix or breast.
  * Acceptable liver, renal, hematologic and coagulation function.

Exclusion Criteria:

* Hematologic malignancies or multiple myeloma.
* For the Dose Expansion cohorts the following cancers are not permitted:

  * Any of the following pure histologies of ovarian cancer: germ cell, sex cord stroma, carcinosarcoma, or sarcoma.
  * Small cell or pure neuroendocrine prostate carcinoma that has not yet been treated with at least one line of platinum-based chemotherapy (prostate adenocarcinoma with immunohistochemical neuroendocrine differentiation but without histological small cell that is naïve to platinum-based chemotherapy will be allowed.)
  * Inflammatory breast cancer.
* New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months, or unstable arrhythmia.
* Cardiac function:

  * Known ejection fraction of <50% by gated radionuclide study (e.g., multi-gated acquisition scan);
  * Fridericia-corrected QT interval (QTcF) >470 msec (female) or >450 msec (male), or history of congenital long QT syndrome;
  * Any ECG abnormality, including pericarditis, that in the Investigator's opinion, would preclude safe participation in the study.
* Active, uncontrolled bacterial, viral, or fungal infections within 7 days of study entry requiring systemic therapy.
* Active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy (thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Known clinically important respiratory impairment.

  * History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
  * History of interstitial lung disease.
* Clinically significant gastrointestinal disorders, such as perforation, gastrointestinal bleeding, or diverticulitis.
* Known to be human immunodeficiency virus (HIV) positive or have hepatitis B surface antigen (HBSAg) or hepatitis C antibodies (HCAb) unless hepatitis C virus (HCV) RNA is undetected/negative.
* History of major organ transplant (i.e., heart, lungs, liver, and kidney).
* History of an allogeneic bone marrow transplant.
* History of an autologous bone marrow transplant within 90 days of study entry.
* Symptomatic central nervous system (CNS) malignancy or metastasis. Patients with treated CNS metastases are eligible, provided their disease is radiographically stable, asymptomatic, and they are not currently receiving corticosteroids and/or anticonvulsants. Radiation must have been completed at least 14 days prior to study entry. Screening of asymptomatic patients without a history of CNS metastases is not required.
* Serious nonmalignant disease that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.
* Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-07-14 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Phase 1b: Number of subjects with dose limiting toxicities which will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE v5.0) | Baseline through 30 days post last dose (5 months)
Phase 1b: Identify the recommended Phase 2 dose (RP2D) of CTX in combination with fixed doses of TRX518 ± avelumab | Baseline through end of Cycle 1 (Day 28)
Phase 2a: Efficacy in Breast and Ovarian Cancer Groups: objective response rate | Baseline to study completion (approximately 4 months)
  To determine the objective response rate according to modified RECIST v1.1
Phase 2a: Efficacy in Prostate Cancer Group: objective response rate | Baseline to study completion (approximately 4 months)
  To determine the objective response rate according to modified RECIST 1.1 and PCWG3 guidelines

SECONDARY OUTCOMES:
To determine the objective disease control rate (ODCR) according to modified RECIST 1.1 in breast and ovarian cancer groups | Baseline to study completion (approximately 4 months)
To determine the objective disease control rate (ODCR) according to modified RECIST 1.1 and PCWG3 guidelines in prostate cancer group | Baseline to study completion (approximately 4 months)
To determine the duration of response according to modified RECIST 1.1 in breast and ovarian cancer groups | Baseline to study completion (approximately 4 months)
To determine the duration of response according to modified RECIST 1.1 and PCWG criteria in prostate cancer group | Baseline to study completion (approximately 4 months)
To determine the progression free survival according to RECIST 1.1 in breast and ovarian cancer groups | Baseline to study completion (approximately 4 months)
To determine the progression free survival according to RECIST 1.1 and PCWG3 criteria in prostate cancer group | Baseline to study completion (approximately 4 months)
To determine overall survival (OS) in all cancer groups | Baseline to study completion (approximately 4 months)
To determine the PSA response in prostate cancer group | Baseline to study completion (approximately 4 months)
Evaluate the effect of TRX518 in combination with cyclophosphamide and avelumab on lymphoid cell subset numbers and function | Various timepoints through study completion (approximately 4 months)
Time to peak concentration (Tmax) | Various timepoints through study completion (approximately 4 months)
  Observations of the distribution, duration of effects and chemical changes of TRX518 and avelumab in the body and the effects and routes of the body's elimination of TRX518 and avelumab
TRX518 and avelumab peak concentration (Cmax) | Various timepoints through study completion (approximately 4 months)
  Observations of the distribution, duration of effects and chemical changes of TRX518 and avelumab in the body and the effects and routes of the body's elimination of TRX518 and avelumab
Area under the curve (AUC) | Various timepoints through study completion (approximately 4 months)
  Observations of the distribution, duration of effects and chemical changes of TRX518 and avelumab in the body and the effects and routes of the body's elimination of TRX518 and avelumab
Assess TRX518 and avelumab immunogenicity | Various timepoints through study completion (approximately 4 months)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Horizon Oncology Research, Lafayette, Indiana
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Virginia, Charlottesville, Virginia